CLINICAL TRIAL: NCT04325035
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study on the Safety and Efficacy of Istaroxime for Pre-Cardiogenic Shock (SEISMiC)
Brief Title: The Safety and Efficacy of Istaroxime for Pre-Cardiogenic Shock
Acronym: SEISMiC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Windtree Therapeutics (Industry)
Collaborators: Momentum Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04-CL-1904; 2020-000885-40 (EudraCT Number)
Record Dates: First submitted 2020-03-24; First posted 2020-03-27 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Cardiogenic Shock
Keywords: Pre-cardiogenic shock; Heart failure
MeSH Terms: conditions — Shock, Cardiogenic; Heart Failure | interventions — Istaroxime

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Matching Placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Istaroxime - Part A (Experimental): Istaroxime IV infusion for 24 hours. Istaroxime administration can begin at 1.0 or 1.5 µg/kg/min; the target infusion rate is 1.5 µg/kg/min
  Interventions: Drug: Istaroxime
- Placebo - Part A (Placebo Comparator): Placebo (lactose lyophilized powder) IV infusion for 24 hours
  Interventions: Drug: Placebo
- Istaroxime - Part B (Experimental): Istaroxime IV infusion at 1.0 µg/kg/min for 6 hours, 0.5 µg/kg/min for 42 hours, 0.25 µg/kg/min for 12 hours.
  Interventions: Drug: Istaroxime
- Istaroxime and Placebo - Part B (Experimental): Istaroxime IV infusion at 0.5 µg/kg/min for 48 hours, followed by placebo IV infusion for 12 hours.
  Interventions: Drug: Istaroxime; Drug: Placebo
- Placebo - Part B (Placebo Comparator): Placebo (lactose lyophilized powder) IV infusion for 60 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Istaroxime — Reconstituted istaroxime and lactose lyophilized powder delivered via IV infusion
  Other Names: PST2744
  Arms: Istaroxime - Part A; Istaroxime - Part B; Istaroxime and Placebo - Part B
Drug: Placebo — Reconstituted placebo (lactose lyophilized powder) delivered via IV infusion
  Other Names: Lactose lyophilized powder
  Arms: Istaroxime and Placebo - Part B; Placebo - Part A; Placebo - Part B

SUMMARY:
This is a pilot, multinational, randomized, double-blind, placebo-controlled, 2-part safety and efficacy study. Subjects will consist of patients hospitalized for acute decompensated heart failure with persistent hypotension.

DETAILED DESCRIPTION:
This is a pilot, multinational, multicenter, randomized, double-blind, placebo-controlled, 2-part safety and efficacy study. Subjects will consist of males or females 18 to 85 years of age, hospitalized for acute decompensated heart failure (ADHF) with persistent hypotension (systolic blood pressure [SBP] 70-100 mmHg for two hours).

Part A will dose all subjects for 24 hours with either 1.0 µg/kg/min or placebo; Part B will dose all subjects for 60 hours with two different regimens of istaroxime or placebo. Enrollment of Part A and Part B will be sequential.

Up to 30 sites in Part A; up to 15 sites in Part B. Sites may be located in Europe, Asia, South America, and North America.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical presentation consistent with SCAI Stage B pre-cardiogenic shock caused by acute decompensation of chronic systolic heart failure (due to arterial hypertension, ischemic heart disease or dilated cardiomyopathy), without evidence for an acute coronary syndrome.
2. Signed informed consent form (ICF);
3. Males and females, 18 to 85 years of age (inclusive);
4. An admission for acute decompensated heart failure (ADHF) episode within 36 hours prior to randomization, defined as:

   1. Dyspnea, at rest or with minimal exertion;
   2. Congestion on chest x-ray or lung US with B-type natriuretic peptide (BNP) ≥ 400 pg/mL or NT-proBNP ≥ 1400 pg/mL; Elective admissions for medications tune up or procedures do not qualify as an ADHF admission.
5. History of left ventricular ejection fraction (LVEF) ≤ 40%;
6. Persistent hypotension defined as:

   1. SBP of 75 to 90 mmHg (Part A) or 70 to 100 mmHg (Part B) for ≥ 2 hours prior to Screening;
   2. SBP does not decrease by > 7 mmHg on two separate measurements during the last 2 hours prior to randomization;
7. Heart rate 75 to 150 bpm. If the subject is on a beta-blocker, the range is 60 to 150 bpm;
8. Echocardiogram during initial hospitalization confirming ejection fraction ≤ 40% and no evidence of other pathology to confound interpretation of cardiac physiology (e.g., pericardial effusion);
9. Subject is monitored by a Pulmonary Artery Catheter (PAC) at the time of randomization (Part B only).

Exclusion Criteria:

1. Cardiogenic shock of SCAI Stage C or worse
2. Cardiogenic shock due to any other condition besides acute decompensation of chronic heart failure.
3. Any of the following in the past 30 days: acute coronary syndrome, coronary revascularization, myocardial infarction (MI), coronary artery bypass graft (CABG), or percutaneous coronary intervention;
4. Current (within 6 hours of Screening) or anticipated need for treatment with positive inotropic agents or vasopressors, renal support including ultrafiltration, or mechanical circulatory, ventilatory or renal support (intra-aortic balloon pump, endotracheal intubation, mechanical ventilation, or any ventricular assist device);
5. Venous Lactate > 2 mmol/L;
6. History of heart transplant or United Network for Organ Sharing (UNOS) priority 1a heart transplant listing
7. Ongoing treatment with digoxin (if digoxin was stopped before signing the ICF and the digoxin plasma level is < 0.5 ng/ml, the patient may be enrolled);
8. Severe renal impairment (estimated glomerular filtration rate (eGFR) < 30 ml/min, calculated by the Modification of Diet in Renal Disease (MDRD) formula);
9. Hypersensitivity to the study medication or any of its excipients (including known lactose hypersensitivity) or any related medication;
10. Stroke or transient ischemic attack (TIA) within 3 months;
11. Active coronary ischemia;
12. Any significant valvular disease (including any moderate or severe valvular stenosis, moderate or severe aortic or pulmonary regurgitation, stenosis or regurgitation);severe tricuspid or mitral regurgitation);
13. Primary hypertrophic or restrictive cardiomyopathy or systemic illness known to be associated with infiltrative heart disease;
14. Admission for AHF triggered primarily by a correctable etiology such as significant arrhythmia, (inclusive of atrial fibrillation as the main reason for admission), infection, severe anemia, acute coronary syndrome, pulmonary embolism, exacerbation of chronic obstructive pulmonary disease (COPD), planned admission for device implantation, or over-diuresis as a cause of hypotension;
15. Pericardial constriction or active pericarditis;
16. Life-threatening ventricular arrhythmia or implantable cardioverter defibrillator (ICD) shock within the past month or history of sudden death within 6 months;
17. Cardiac resynchronization therapy (CRT), ICD, or pacemaker implantation (or planned implantation) within the past 3 months;
18. Sustained ventricular tachycardia in the last 3 months with no defibrillator;
19. Sustained hypotension (SBP < 70 mmHg) for at least 30 minutes from the time of arrival to the hospital;
20. Severe pulmonary disease or cor pulmonale or other causes of isolated right-sided HF or not related to left ventricular dysfunction;
21. Acute respiratory distress syndrome;
22. Suspected sepsis; fever > 38°C or active infection requiring IV antimicrobial treatment;
23. Body weight < 40 kg or ≥ 150 kg;
24. Laboratory exclusions:

    1. Hemoglobin < 9 g/dl,
    2. Platelet count < 100,000/µl,
    3. Serum potassium > 5.3 mmol/l or < 3.5 mmol/l;
25. A life expectancy < 3 months based on the judgment of the investigator;
26. Uncontrolled thyroid disease;
27. Pregnant or breast-feeding;
28. Ongoing drug or alcohol abuse;
29. Participation in another interventional study within the past 30 days.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in systolic blood pressure (SBP) area under the curve (AUC) 0-6 | 0 to 6 hours after initiation of infusion
  Change from baseline AUC for systolic blood pressure

SECONDARY OUTCOMES:
Change from baseline in SBP AUC 0-48 | 0 to 60 hours after initiation of infusion
  Change from baseline in AUC for systolic blood pressure in Part B
Change from baseline in SBP AUC 0-60 | 0 to 48 hours after initiation of infusion
  Change from baseline in AUC for systolic blood pressure in Part B
Treatment failure score | 60 hours from initiation of infusion
  Treatment-failure score, based on death, circulatory, respiratory, or renal mechanical support or intravenous inotrope or vasopressor treatment, and changes in systolic blood pressure
Change from baseline in SBP | 6 hours after initiation of infusion
  Change from baseline in systolic blood pressure
Change from baseline in SBP | 24 hours after initiation of infusion
  Change from baseline in systolic blood pressure
Change from baseline in SBP | 48 hours after initiation of infusion
  Change from baseline in systolic blood pressure in Part B
Change from baseline in SBP | 60 hours after initiation of infusion
  Change from baseline in systolic blood pressure in Part B
Number of treatment failures | Randomization to 24 hours for Part A
  Number of subjects requiring treatment with intravenous vasopressors, inotropes, and/or mechanical cardiac or renal support or have died
Number of treatment failures | Randomization to 48 hours for Part B
  Number of subjects requiring treatment with intravenous vasopressors, inotropes, and/or mechanical cardiac or renal support or have died
Number of treatment failures | Randomization to Day 5
  Number of subjects requiring treatment with intravenous vasopressors, inotropes, and/or mechanical cardiac or renal support or have died
Change in quality of life | Baseline to Day 5 (96 hours) from infusion start
  Changes from baseline measured by the EQ-5D in Part A
Change in quality of life | Baseline to Day 30 from infusion start
  Changes from baseline measured by the EQ-5D in Part A
Change in eGFR | 24 hours from infusion start
  Change from baseline and observed estimated glomerular filtration rate (eGFR)
Change in eGFR | 48 hours from infusion start
  Change from baseline and observed estimated glomerular filtration rate (eGFR)
Change in brain natriuretic peptide (BNP), N-terminal pro hormone B-type natriuretic peptide (NT-pro-BNP), troponin (cTn; either T or I) and venous lactate | 24 hours from infusion start
  Change from baseline and observed BNP, NT-pro-BNP, troponin (cTn; either T or I) and venous lactate
Change in brain natriuretic peptide (BNP), N-terminal pro hormone B-type natriuretic peptide (NT-pro-BNP), troponin (cTn; either T or I) and venous lactate | 48 hours from infusion start
  Change from baseline and observed BNP, NT-pro-BNP, troponin (cTn; either T or I) and venous lactate
Time to worsening heart failure (HF) | Up to Day 5
  Time to worsening HF
Time to HF re-admission or death | Up to Day 30
  Time to HF re-admission or death
Length of initial hospitalization | Up to Day 30
  Length of initial hospitalization
Days alive and out of the hospital | Up to Day 30
  Days alive and out of the hospital
Mortality and reasons for death | Up to Day 30
  Mortality and reasons for death
Change in coronary index (CI) | 24 hours
  Change from baseline in CI as assessed by echocardiogram - Part A
Change in E to e' ratio | 24 hours
  Change from baseline in E to e' ratio as assessed by echocardiogram - Part A
Change in stroke volume index (SVI) | 24 hours
  Change from baseline in SVI as assessed by echocardiogram - Part A
Change in left atrium area (LAA) | 24 hours
  Change from baseline in LAA as assessed by echocardiogram - Part A
Change in CI | 48 hours
  Change from baseline in CI as assessed by echocardiogram - Part B
Change in E to e' ratio | 48 hours
  Change from baseline in E to e' ratio as assessed by echocardiogram - Part B
Change in SVI | 48 hours
  Change from baseline in SVI as assessed by echocardiogram - Part B
Change in LAA | 48 hours
  Change from baseline in LAA as assessed by echocardiogram - Part B

CONTACTS AND LOCATIONS:
Overall Officials: Marco Metra, MD, Principal Investigator — Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia, Italy
Locations (13):
- Tufts Medical Center, Boston, Massachusetts, United States
- Argentina (5):
  - Hospital Italiano de Bueno Aires, Capital Federal, Buenos Aires
  - Santorio Guemes, Capital Federal, Buenos Aires
  - Hospital Privado de Rosario, Rosario, Sante Fe
  - Instituto Cardiovascular de Rosario, Rosario, Sante Fe
  - Santorio de la Trinidad Palermo, Buenos Aires
- Italy (3):
  - Azienda Ospedaliera Santi Antonio e Biagio e Cesare Arrigo, Alessandria
  - UOC Cardiologia, ASST degli Spedali Civili di Brescia Pizzale Spedali Civili 1, Brescia
  - IRCCS San Raffaele Scientific Institute, Milan
- Poland (4):
  - Uniwersytecki Szpital Kliniczny, Centrum Chorub Serca, Wroclaw, Lower Silesian Voivodeship
  - Uniwersytecki Szpital Kliniczny w Białymstoku, Bialystok
  - Uniwersytecki Szpital Kliniczny w Opolu, Opole
  - 4 Wojskowy Szpital Kliniczny, Wroclaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Metra M, Chioncel O, Cotter G, Davison B, Filippatos G, Mebazaa A, Novosadova M, Ponikowski P, Simmons P, Soffer J, Simonson S. Safety and efficacy of istaroxime in patients with acute heart failure-related pre-cardiogenic shock - a multicentre, randomized, double-blind, placebo-controlled, parallel group study (SEISMiC). Eur J Heart Fail. 2022 Oct;24(10):1967-1977. doi: 10.1002/ejhf.2629. Epub 2022 Aug 22. PMID 35867804
- [Result] Metra M, Chioncel O, Davison B, Filippatos G, Mebazaa A, Pagnesi M, Adamo M, Novosadova M, Ponikowski P, Simmons P, Soffer J, Simonson S, Cotter G. Safety and Efficacy of Istaroxime 1.0 and 1.5 microg/kg/min for Patients With Pre-Cardiogenic Shock. J Card Fail. 2023 Jul;29(7):1097-1103. doi: 10.1016/j.cardfail.2023.03.020. Epub 2023 Apr 17. PMID 37075941